CLINICAL TRIAL: NCT05706831
Title: Music Intervention and Transcranial Electrical Stimulation for Treating Neurological Diseases
Brief Title: Music Intervention and Transcranial Electrical Stimulation for Neurological Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Bari Aldo Moro (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Simona Spaccavento, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 345
Record Dates: First submitted 2022-11-16; First posted 2023-01-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Disorder of Consciousness; Stroke
Keywords: music stimulation; tDCS; Aphasia; Neglect; DOC; Stroke
MeSH Terms: conditions — Consciousness Disorders; Stroke; Aphasia

STUDY DESIGN:
Intervention Model Description: Three groups of neurological patients will be considered for the study. For each group, participants will be randomly allocated to one of three intervention groups. These interventions will consist of a combination of musical stimulation, sham stimulation, tDCS and noise.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Group 1 will receive tEs combined with music stimulation for 2 weeks, 1 week of wash out, then sham stimulation combined with noise (placebo) for other 2 weeks.
  Interventions: Other: Combinatory effect of music stimulation and neurostimulation
- Group 2 (Experimental): Group 2 will receive sham stimulation and noise (placebo) for the first 2 weeks, then 1 week wash out, and finally tEs and music stimulation for other 2 weeks.
  Interventions: Other: Combinatory effect of music stimulation and neurostimulation
- Group 3 (Experimental): Group 3 will receive only music stimulation and sham stimulation for 2 weeks, 1 week of wash out, then sham stimulation and noise (placebo) for another 2 weeks.
  Interventions: Other: Combinatory effect of music stimulation and neurostimulation

INTERVENTIONS:
Other: Combinatory effect of music stimulation and neurostimulation — music

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a musical interventionand non-invasive brain stimulation in neurological patients. The main questions it aims to answer are:

* to evaluate the residual neuroplastic processes in DOC state related to music exposure
* to determine the putative modulation of the aforementioned processes and the clinical outcome of DOC patients by non-pharmacological strategies, i.e., electric (tDCS) and music stimulation
* to evaluate the impact of this intervention on caregiver's burden and psychological distress.

Participants will be randomly assigned to one of three different music-listening intervention groups. Primary outcomes will be clinical, that is based on the neurologist's observations of clinical improvement, and neurophysiological, collected pre-intervention, post-intervention and post-placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Post-stroke aphasia
* Post-stroke neglect
* Patients with disorders of consciusness (DOC)

Exclusion Criteria:

* No auditory injury
* no hystory of neurological disease
* No hystory of psychiatric disease
* Previous stroke
* use of alcohol and drugs
* premorbid dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological outcomes | Change from baseline Coma Recovery Scale- Revised at 2 weeks and 4 weeks
  -Coma Recovery Scale-Revised (CRS-R) - (0-23). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Disability Rating Scale at 2 weeks and 4 weeks
  Disability Rating Scale (DRS) - (0-29). High score means a worse outcome.
Neuropsychological outcomes | Change from baseline Rancho Levels of Cognitive Functioning at 2 weeks and 4 weeks
  Rancho Levels of Cognitive Functioning (LCF) - (1-8). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Glasgow Outcome Scale- Extended at 2 weeks and 4 weeks
  Glasgow Outcome Scale- Extended (GOS-E) - (1-8). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Aachener Aphasie Test at 2 weeks and 4 weeks
  Aachener Aphasie Test (AAT). This test includes six subtests: spontaneous speech, token test, repetition, written language, naming, and comprehension.
  Spontaneous speech is structured in six parts (0-30). High score means a better performance; Token test is composed by 50 items; for the score the number of error id considered (0-50).
  Repetition sub test is composed by 50 items; for each item the score range from 0 to 3; high score means better outcome (0-150).
  Written language subtest is composed by 30 items; for each item the score range from 0 to 3; high score means better outcome (0-90).
  Naming subtest is composed by 40 items; for each item the score range from 0 to 3; high score means better outcome (0-120).
  Comprehension subtest is composed by 40 items; for each item the score range from 0 to 3; high score means better outcome (0-120).
Neuropsychological outcomes | Change from baseline Italian version of Functional Outcome Questionnaire for Aphasie at 2 weeks and 4 weeks
  Italian version of Functional Outcome Questionnaire for Aphasie (FOQ-A) - (32-160). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Functional Assessment Measure - Cognitive subscale at 2 weeks and 4 weeks
  Functional Assessment Measure - Cognitive subscale - (FAM) - (14-98); high score means a better outcome.
Neuropsychological outcomes | Change from baseline Quality of Life Questionnaire for aphasics at 2 weeks and 4 weeks
  Quality of Life questionnaire for Aphasics (QLQA) - (0-148); High score means a better outcome.
Neuropsychological outcomes | Change from baseline The semi-structured scale for functional evaluation of personal neglect at 2 weeks and 4 weeks
  The semi-structured scale for functional evaluation of personal neglect - (0-9); High score means a worse outcome.
Neuropsychological outcomes | Change from baseline Barrage Test at 2 weeks and 4 weeks
  Barrage test (0-36). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Letter cancellation test at 2 weeks and 4 weeks
  Letter cancellation test - (0-104). High score means a better outcome.
Neuropsychological outcomes | Change from baseline Sentence reading test at 2 weeks and 4 weeks
  Sentence reading test (0-6). High score means a worse outcome.
Neuropsychological outcomes | Change from baseline Wundt-Jastrow area illusion test at 2 weeks and 4 weeks
  Wundt-Jastrow area illusion test (0-20). High score means a worse outcome.
Neuropsychological outcomes | Change from baseline The semi structured scale for the functional evaluation of extrapersonal neglect at 2 weeks and 4 weeks
  The semi structured scale for the functional evaluation of extrapersonal neglect (0-9). High score means a worse outcome.
Neurophysiological outcome | Change from baseline oscillation at 2 weeks and 4 weeks
  The ratio of fast (8-30 Hz, α-β) to slow (2-8 Hz, δ-θ) oscillation amplitude at the midline electrodes (Fz, Cz, Pz, Oz) will be measured and compared pre- and post intervention."

SECONDARY OUTCOMES:
Caregiver psychological distress | Change from baseline Back depression Inventory II at 2 weeks and 4 weeks
  Back depression Inventory II (BDI II) - (0-63). High score means a worse outcome.
Caregiver psychological distress | Change from baseline State-trait anxiety inventory; at 2 weeks and 4 weeks
  State-trait anxiety inventory (STAI-Y). It is composed by two scales: STAI-Y State (20-80) and STAI-Y Trait (20-80). High score means a worse outcome.
Caregiver psychological distress | Change from baseline Questionario psicofisiologico (CBA) at 2 weeks and 4 weeks
  Psychophysiological Questionnaire (30-120). WHOQOL-BREF.
Caregiver psychological distress | Change from baseline Prolonged grief disorder -12 at 2 weeks and 4 weeks
  Prolonged grief disorder -12 (PG-12) - (11-55). High score means a worse outcome.
Caregiver psychological distress | Change from baseline Family strain questionnaire at 2 weeks and 4 weeks
  Family strain questionnaire (FSQ) - (1-44). High score means a worse outcome.
Caregiver psychological distress | Change from baseline Wolrd health organization - quality of life at 2 weeks and 4 weeks
  better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Bari, Ba, Italy

REFERENCES:
- [Derived] Spaccavento S, Carraturo G, Brattico E, Matarrelli B, Rivolta D, Montenegro F, Picciola E, Haumann NT, Jespersen KV, Vuust P, Losavio E. Musical and electrical stimulation as intervention in disorder of consciousness (DOC) patients: A randomised cross-over trial. PLoS One. 2024 May 31;19(5):e0304642. doi: 10.1371/journal.pone.0304642. eCollection 2024. PMID 38820520